CLINICAL TRIAL: NCT04779554
Title: A Randomized Phase 2 Trial of Flat Dose vs. Weight-based Dose of Intra-peritoneal (IP) Chemotherapy for Patients Undergoing Cytoreductive Surgery and Heated Intra-peritoneal Chemotherapy (CRS/HIPEC) for Advanced Gastrointestinal Malignancy
Brief Title: Flat Dose vs. Weight-based IP Chemotherapy for CRS/HIPEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prakash Pandalai (Other)
Responsible Party: Sponsor-Investigator, Prakash Pandalai, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GI-115
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal Carcinomatosis
Keywords: cytoreductive surgery; colorectal cancer; pseudomyxoma peritonei; appendiceal mucinous neoplasm; mitomycin C; pharmacokinetics; CRS/HIPEC; HIPEC; Appendix cancer; LAMN
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms; Pseudomyxoma Peritonei; Appendiceal Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Flat Dose Mitomycin C (Experimental): Participants in this group will receive flat doses of mitomycin C intra-operatively: 1) 30mg at minute 0 and 2) 10mg at minute 45. Mitomycin C will be delivered via HIPEC (hyperthermic intraperitoneal chemotherapy).
  Interventions: Drug: Mitomycin C, flat dose 40 mg
- Weight-Based Mitomycin C (Experimental): Participants in this group will receive weight-based dosing of mitomycin C intra-operatively: 1) 9.5 mg/m2 at minute 0 and 2) 3 mg/m2 at minute 45 for total dose of 12.5 mg/m2. Mitomycin C will be delivered via HIPEC (hyperthermic intraperitoneal chemotherapy).
  Interventions: Drug: Mitomycin C, weight-based dose 12.5 mg/m2

INTERVENTIONS:
Drug: Mitomycin C, flat dose 40 mg — Mitomycin C will be delivered as heated intraperitoneal chemotherapy (HIPEC) in two flat doses. Dose 1 will be 30mg at minute 0 and dose 2 will be 10 mg at minute 45.
  Arms: Flat Dose Mitomycin C
Drug: Mitomycin C, weight-based dose 12.5 mg/m2 — Mitomycin C will be delivered as heated intraperitoneal chemotherapy (HIPEC) in two weight-based doses of 9.5 mg/m2 at minute 0 and 3 mg/m2 at minute 45.
  Arms: Weight-Based Mitomycin C

SUMMARY:
Peritoneal carcinomatosis from advanced gastro-intestinal malignancy has historically been associated with poor overall survival (≤ 12 months) with few treatment options. Cytoreductive surgery (CRS), which involves removal of all macroscopic tumor nodules, combined with direct administration of heated intra-peritoneal (IP) chemotherapy (HIPEC) to the affected peritoneal surfaces, has been shown to be an effective treatment option that extends overall survival among certain cases of peritoneal carcinomatosis. IP chemotherapy allows delivery of a high dose of cytostatic drug directly onto the peritoneal surfaces at risk for microscopic residual disease while systemic exposure remains limited. Additionally, hyperthermia is known to enhance the cytotoxicity of several agents (including Mitomycin C) and improves the depth of peritoneal penetration.

This trial will be a randomized phase 2 comparison of flat dose versus weight-based dose Mitomycin C. The hypothesis of this study is that HIPEC weight-based dosing may result in similarly effective peritoneal Mitomycin C concentrations with less systemic absorption and potential systemic toxicity, compared with the HIPEC flat dosing approach in patients undergoing CRS/HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with one of the following: low-grade appendiceal mucinous neoplasm, pseudomyxoma peritonei, appendiceal cancer with peritoneal carcinomatosis, colorectal cancer with peritoneal carcinomatosis
* ECOG performance status < 3
* Candidate for grossly complete cytoreductive surgery
* Life expectancy greater than 3 months
* Adequate organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any extra-abdominal metastases
* Untreated lung metastases
* Liver metastases not amenable to resection or ablation
* Known brain metastases
* Chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Presence of residual significant adverse events attributed to prior cancer treatment
* Currently receiving any other investigational therapeutic agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Mitomycin C.
* Pregnant or breast-feeding women
* Uncontrolled ongoing illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) - Pharmacokinetics | Approximately 20 hours
  Drug exposure will be measured by calculating the area under the curve (AUC) or integral of a plasma concentration-time curve. Samples will be collected at 0,15, 30, 60 and 90 minutes intra-operatively, and 2, 4, and 12 hours postoperatively.
Drug Clearance (CL) - Pharmacokinetics | Approximately 20 hours
  Drug clearance will be calculated as the volume of plasma cleared per unit time. Samples will be collected at 0,15, 30, 60 and 90 minutes intra-operatively, and 2, 4, and 12 hours postoperatively.
Drug Half-Life (T1/2) - Pharmacokinetics | Approximately 20 hours
  Drug half-life will be calculated as the time required for the plasma Mitomycin C concentration to be half of its maximum concentration. Samples will be collected at 0,15, 30, 60 and 90 minutes intra-operatively, and 2, 4, and 12 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Pandalai, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald HG, Cassim EB, Harper MM, Burke EE, Marcinkowski EF, Cavnar MJ, Pandalai PK, Kim J. The Development of Investigator-Initiated Clinical Trials in Surgical Oncology. Surg Oncol Clin N Am. 2023 Jan;32(1):13-25. doi: 10.1016/j.soc.2022.07.003. Epub 2022 Nov 3. PMID 36410913